CLINICAL TRIAL: NCT00676429
Title: Ziprasidone for Severe Conduct and Other Disruptive Behavior Disorders in Children and Adolescents - a Placebo Controlled, Randomized, Double Blind Clinical Trial
Brief Title: Ziprasidone for Severe Conduct and Other Disruptive Behavior Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Professor Dr. Eberhard Schulz, MD, University Hospital Freiburg, Dept. of Child & Adolescent Psychiatry
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRA1280023; EudraCT: 2006-002207-13
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2008-11-18 (Estimated); Status verified 2008-11

CONDITIONS: Conduct Disorder; Oppositional Defiant Disorder
MeSH Terms: conditions — Conduct Disorder; Oppositional Defiant Disorder | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Ziprasidone Hydrochloride oral solution with individual titration from 5 mg to 40 mg per day
  Interventions: Drug: Ziprasidone Hydrochloride
- 2 (Placebo Comparator): Placebo oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ziprasidone Hydrochloride — Ziprasidone Hydrochloride oral solution, individual titration 5 mg o.d. or 10 mg to 40 mg b.i.d
  Other Names: Zeldox 10mg/ml Suspension zum Einnehmen
  Arms: 1
Drug: Placebo — Placebo as oral solution, individually titrated
  Other Names: Placebo Suspension zum Einnehmen
  Arms: 2

SUMMARY:
To investigate and compare the efficacy, safety and tolerability of ziprasidone versus placebo in the treatment of conduct disorder (CD), oppositional defiant disorder (ODD) and disruptive behavior disorder not otherwise specified (DBD-NOS) of older children and adolescents in an outpatient setting.

Conduct and other behavior disorders are some of the most common forms of psychopathology in children and adolescents. The main characteristic of these disorders is a repetitive and persistent pattern of antisocial, aggressive or defiant behavior that involves major violations of age-appropriate expectations or norms. According to the guidelines of the German Society for Child & Adolescent Psychiatry & Psychotherapy (Deutsche Gesellschaft für Kinder- und Jugendpsychiatrie und -psychotherapie DGKJPP), the European Society for Child and Adolescent Psychiatry (ESCAP), and the American Academy of Child and Adolescent Psychiatry (AACAP) currently no standard pharmacotherapy is established and recommended for children and adolescents. However Risperidone has been shown to be effective in the treatment of patients with disruptive behavior disorders and below average IQ.

DETAILED DESCRIPTION:
Trial Design:

A placebo-controlled, parallel-group, randomized, double-blind, single center design that includes a 3-weekly baseline period for finding the best individual dose, a 6-weeks treatment period and a 2-weeks washout period.

Study Agent / Placebo - Dosage and Route of Administration:

Study medication will first be dispensed at Visit 2 (day 1). Treatment assignments will be made in accordance with the randomization sequence. At each medication visit (Visit 2 to Visit 7), subjects will receive one bottle for the following week (Visit 2 to Visit 4) resp. the following two weeks (Visit 5 to Visit 7). Only qualified personnel may dispense study medication.

The study population will be randomized equally to the verum or placebo group at Visit 2. All patients will receive an initial oral course starting with 5mg/d Ziprasidone Hydrochloride or placebo for patients with a body weight ≤ 50 kg and 10 mg/d Ziprasidone Hydrochloride or placebo for patients with a body weight > 50 kg for the first week in the study.

At Visit 3 the therapist can increase the dose to the double of the initial dose according to clinical response and tolerability. At Visit 4 the dose can be increased to the double of the last dose or reduced to the initial dose. At Visit 5 the most effective and best tolerated dose will be given for the 6 week fixed dose phase of the trial. Therefore the maximum daily dose is 20 mg (patients with body weight ≤ 50 kg) or 40 mg (patients with body weight > 50 kg). The total dose will be split and the half-dose will be given twice a day (morning and evening).

Planned Study Time Schedule:

The study ends 11 weeks after enrollment of the last patient (total study end). Study duration for each patient is 11 weeks (from inclusion) until the last visit (close-out visit). Patients with a pre-treatment of psychotropic drugs will have an individual washout period before inclusion to the study. This individual washout period will last 5 elimination half-life of the taken drug.

After randomization the patients will enter a 3 week dose escalation phase with weekly visits. Then a 6 week stable drug dose phase will follow with visits every second week, followed by a two week washout period and a final visit.

Statistics:

Sample size calculation:

Sample size calculation is based on the assumption that treatment with Ziprasidone will show an effect size of ES=1 compared to treatment with placebo. In order to demonstrate this difference at a significance level of 5% and a power of 80%, 17 patients per group are required, and a drop-out rate of approximately 8 patients per group (with no data available to be analyzed according to the intention-to-treat principle) must be accounted for.

Analysis of efficacy:

The trial will be analyzed according to the intention-to-treat principle. The effect of treatment with Ziprasidone will be assessed by analyzing changes in the score of the scale described above. Changes calculated from the evaluations before and after treatment will be analyzed by means of analysis of covariance, considering the baseline measurement as a covariate. The difference between treatment groups will be estimated with a 95% confidence interval and will be tested within this model by the corresponding two-sided test at the 5% level of significance.

Analysis of safety:

Safety analyses will be performed for patients who received at least one dose of the investigational drug. Rates of adverse events and of serious adverse events will be calculated with corresponding 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* The subject and the authorized legal representative must understand the nature of the study and be able to comply with protocol requirements. The representative must sign an Informed Consent Document and the subject must provide Written Assent.
* The subject (male or female) must be between 7-17 (inclusive) years of age at screening.
* The subject must have a primary diagnosis of Conduct Disorder [CD] (312.8), Oppositional Defiant Disorder [ODD] (313.81) or Disruptive Behavior Disorder not otherwise specified [DBD-NOS] (312.9) as defined by DSM-IV criteria and confirmed by the Kiddie-SADS-PL.
* At the screening visit (Visit 1), subjects must have a score of 21 or more on the sum of the scales for conduct problems and for oppositional behaviour in the NCBRF-TIQ.
* In the investigator's opinion, the subject must be likely to benefit from the therapy.
* The subject is willing and able to discontinue any medications that are prohibited in this study (see Concomitant Medications table, Section 3.5.1). Any such medications must be discontinued at least 5 half-lives prior to the administration of double-blinded study medication.
* Patients who are receiving prohibited medications are to be considered for the protocol only If discontinuation of the medication does not compromise the welfare of the patient and/or alternative medication that is allowed by the protocol is available and appropriate for the patient. Psychotropic medications should be tapered down per accepted medical practice and the specific package insert instead of being abruptly discontinued.
* Females of childbearing potential may be included provided that they are not pregnant, not nursing, and are practicing effective contraception and meet all of the following criteria:

  * Are instructed and agree to avoid pregnancy during the study.
  * Have a negative pregnancy test (β-HCG) at screening and Visit 2.
  * Use one of the following birth control methods:

    * an oral contraceptive agent, an intrauterine device (ILTD), an implantable contraceptive (e.g. Norplant), transdermal hormonal contraceptive (e.g. Ortho-Evra), or an injectable contraceptive (e.g. Depo-Provera) for at least one month prior to entering the study and will continue its use throughout the study; or
    * a barrier method of contraception, e.g., condom and / or diaphragm with spermicide while participating in the study.
    * abstinence for at least 3 months before the start of the study and intention to abstain from sexual activity during the study period.
* Subjects must have an IQ > 55 best tested with the HAWIK-III, alternatively with the CFT-20 or K-ABC.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Nisonger Child Behavior Rating Form for typical IQ (NCBRF-TIQ): Combined subscales "Conduct Problem" and "Oppositional Behavior" | Visit 2 to Visit 9 (week 0, 1, 2, 3, 5, 7, 9 and 11)

SECONDARY OUTCOMES:
Assessment of the safety and tolerability by adverse event documentation. | Visit 2 to Visit 9 (week 0, 1, 2, 3, 5, 7, 9 and 11)
Assessment of the efficacy by the Clinical Global Impressions-Severity of Illness scale (CGI-S) and the Global Impressions-Improvement scale (CGI-I). | Visit 2 to Visit 9 (week 0, 1, 2, 3, 5, 7, 9 and 11)
Correlation between dosage, efficacy and adverse events. | Visit 2 to Visit 9 (week 0, 1, 2, 3, 5, 7, 9 and 11)
Ziprasidone serum levels | Visit 5 (week 3) and Visit 8 (week 8)
Correlation between serum level, efficacy and adverse events | Visit 5 (week 3) and Visit 8 (week 8)

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Schulz, MD, Principal Investigator — University Hospital Freiburg, Dep. for Child & Adolescent Psychiatry; Christian Fleischhaker, MD, Study Chair — University-Hospital Freiburg, Dep. for Child & Adolescent Psychiatry; Klaus Hennighausen, MD, Study Director — University Hospital Freiburg
Locations (1):
- University Hospital Freiburg, Dep. for Child & Adolescent Psychiatry, Freiburg im Breisgau, Germany